CLINICAL TRIAL: NCT01271283
Title: Lenalidomide for the Treatment of CLL Patients With High-Risk Disease
Brief Title: Lenalidomide in Treating Patients With High-Risk Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02568; NCI-2011-02568 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000692070; RPCI # I 174910 (Other: Roswell Park Cancer Institute); 8254 (Other: CTEP); P30CA016056 (NIH)
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

ARMS (1):
- Arm I (Experimental): Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (by morphological criteria but have persistent minimal residual disease by molecular criteria) or partial response may continue treatment beyond 8 courses. Patients may undergo bone marrow, peripheral blood, and/or lymph node sample collection at baseline and periodically during study for correlative studies.
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given orally
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II clinical trial is studying how well lenalidomide works in treating patients with high-risk chronic lymphocytic leukemia. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the time to progression in patients with high-risk chronic lymphocytic leukemia (CLL) treated with lenalidomide.

SECONDARY OBJECTIVES:

I. To determine the clinical response (complete and partial response) in treatment-naïve patients with high-risk CLL treated with single-agent lenalidomide.

II. To determine the incidence of immune-mediated flare reaction. III. To determine the toxicity profile of single-agent lenalidomide in previously untreated patients with high-risk CLL.

IV. To conduct correlative studies in bone marrow, peripheral blood, and/or lymph nodes of patients treated with lenalidomide.

OUTLINE:

Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (by morphological criteria but have persistent minimal residual disease by molecular criteria) or partial response may continue treatment beyond 8 courses. Patients may undergo bone marrow, peripheral blood, and/or lymph node sample collection at baseline and periodically during study for correlative studies.

After completion of study therapy, patients are followed up every 3 months for a maximum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of B-cell chronic lymphocytic leukemia (B-CLL) as defined by the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria

  * Must have high-risk B-CLL as defined by ≥ one of the following:

    * High-risk cytogenetics (either 17p deletion and/or 11q deletion)
    * Unmutated immunoglobulin heavy chain gene rearrangement
  * Zap-70 and CD38 expression on leukemic cells will not be used as eligibility criteria for enrollment into the clinical trial
* No prior treatment for the management of B-CLL
* Patients must have B-CLL requiring therapy as defined by the IWCLL criteria
* Must have measurable disease meeting one of the following criteria:

  * Absolute lymphocyte count > 5,000/μL
  * Measurable lymphadenopathy or organomegaly
* No tumor lysis syndrome (TLS) by Cairo-Bishop definition

  * Patients with correction of electrolyte abnormalities allowed
* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Creatinine clearance ≥ 30 mL/min
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN (≤ 5 times ULN if hepatic metastases are present)
* Uric acid normal

  * Patients with elevated uric acid allowed provided it is corrected with appropriate pharmacologic measures
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must commit to continued abstinence from heterosexual intercourse or use 2 acceptable methods of contraception (1 highly effective method and 1 additional effective method) ≥ 28 days prior to, during, and for ≥ 28 days after discontinuing lenalidomide
* Able to adhere to the study visit schedule and other protocol requirements
* No serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form
* No condition, including the presence of laboratory abnormalities, that would place the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* No known hypersensitivity to thalidomide or lenalidomide
* No history of erythema nodosum characterized by a desquamating rash while taking thalidomide or similar drugs
* No history of any other cancer except non-melanoma skin cancer or carcinoma in-situ of the cervix or cancer for which the patient is in complete remission and off therapy for > 3 years
* No cardiac arrest within the past 6 months
* No known history of hepatitis B infection, positive hepatitis B surface antigen, or positive hepatitis C antibody
* No other concurrent anti-cancer agents or treatments
* More than 28 days since any prior experimental drug or therapy
* Aspirin (81 or 325 mg) or warfarin sodium daily as prophylactic anticoagulation required
* No prior lenalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Time to progression | From the start of lenalidomide therapy to time of disease progression, assessed up to 24 months

SECONDARY OUTCOMES:
Maximal clinical response (complete and partial response) | Up to 24 months
  Summarized by a sample proportion along with the exact 95% confidence interval. The time-to-progression will be graphically analyzed using standard Kaplan-Meier estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Asher Chanan-Khan, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States